CLINICAL TRIAL: NCT04639284
Title: Combination Therapy With Anti-angiogenic Agents and Anti-PD-1 Antibodies for Unresectable or Advanced Hepatocellular Carcinoma: a Cohort Study
Brief Title: Anti-angiogenic Agents Plus Anti-PD-1 Antibodies for uHCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Professor of Surgery, Shanghai Zhongshan Hospital
Other Study IDs: COMOHCC
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: anti-angiogenic; PD-1 antibody; lenvatinib; PD-L1 antibody
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Angiogenesis Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue specimens and blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combinational therapy: Participants who receive systemic treatment with an anti-angiogenic agent, including sorafenib, lenvatinib, apatinib, and bevacizumab, in combination with an anti-PD-1/PD-L1 antibody, including pembrolizumab, nivolumab, sintilimab, toripalimab, camrelizumab, tislelizumab, and atezolizumab.
  Interventions: Drug: Anti-angiogenic agents plus anti-PD-1/PD-L1 antibodies

INTERVENTIONS:
Drug: Anti-angiogenic agents plus anti-PD-1/PD-L1 antibodies — Combination therapies with an anti-angiogenic agent (tyrosine kinase inhibitor or VEGF/VEGFR antibody) and an anti-PD-1/PD-L1 antibody.

SUMMARY:
Combination treatment with antiangiogenic agents and anti-programmed cell death protein 1 (PD-1) antibodies have shown high anti-tumor efficacy for patients with unresectable or advanced hepatocellular carcinoma (uHCC). In this single-center cohort study, we are aiming to (1) evaluate the clinical effectiveness in real-world patients, especially for Chinese patients, most of whom were with hepatitis B virus infection; (2) predict clinical effectiveness with clinicopathological features; (3) predict clinical effectiveness with histologic features and blood samples.

DETAILED DESCRIPTION:
Combination treatment with antiangiogenic agents and anti-programmed cell death protein 1 (PD-1) antibodies have shown high anti-tumor efficacy for patients with unresectable or advanced hepatocellular carcinoma (uHCC). In this single-center cohort study, we are aiming to:

1. To evaluate the clinical effectiveness in real-world patients, especially for Chinese patients most of whom were with hepatitis B virus infection.
2. To predict clinical effectiveness with clinicopathological features, such as lab examinations (at baseline and dynamic changes), radiological features (radiomics study at the baseline);
3. To predict clinical effectiveness with histologic features, such as PD-L1 expression, ctDNA, and peripheral immune cell subtypes.
4. To evaluate the clinical effectiveness of second- or third-line therapies, including TACE, HAIC, and interferon, for those who lost clinical benefit or who were intolerant to the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of HCC confirmed by histology/cytology or clinical diagnosis of HCC by Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2019 edition) criteria.
2. Unresectable or advanced disease at the investigator's discretion. The advanced stage was BCLC C stage or China Liver Cancer Stage IIIa or IIIb.
3. Child-Pugh class A or B7.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Subjects received combination therapy with an anti-angiogenic agent and an anti-PD-1/PD-L1 antibody, received at least one imaging evaluation, and signed an Informed Consent Form. Anti-angiogenic agents include sorafenib, lenvatinib, apatinib, and bevacizumab; anti-PD-1/PD-L1 antibodies include pembrolizumab, nivolumab, sintilimab, toripalimab, camrelizumab, tislelizumab, and atezolizumab.
6. Adequate hematologic and end-organ function.

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
2. History of malignancy other than HCC within 5 years prior to the therapy, with the exception of adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or papillary thyroid carcinoma.
3. History of organ transplantation or hepatic encephalopathy.
4. Allergic to anti-angiogenic agents or anti-PD-1/PD-L1 agents.
5. History of gastrointestinal perforation and/or fistula within the 6 months, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection, Crohn's disease, ulcerative colitis, or chronic diarrhea within 6 months.
6. Active autoimmune disease requiring systemic therapy within 2 years prior to the first dose, allowing the use of alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency); history of primary immunodeficiency; presence of only autoimmune antibody-positive subjects. The presence of autoimmune disease needs to be confirmed at the investigator's discretion.
7. Uncontrollable hypertension, SBP >140 mmHg or DBP >90 mmHg after optimal medical therapy, hypertensive crisis, or history of hypertensive encephalopathy.
8. Subjects had a bleeding event in the past 6 months due to esophageal or gastric fundus varices induced by portal venous hypertension; subjects have undergone a gastrointestinal endoscopy within 3 months prior to the first dose to diagnose the presence of severe (G3) varices; subjects had a high risk of bleeding as assessed by the investigator.
9. Subject requests withdrawal of informed consent.
10. Other conditions that the investigator deems inappropriate for participation in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable or advanced HCC patients who received the combination therapy with an anti-angiogeic agent and an anti-PD-1/PD-L1 agent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response | up to 2 years
  Subjects with complete response or partial response

SECONDARY OUTCOMES:
Duration of response | up to 2 years
  the interval between the time of partial or complete response to the time of progressive disease
Progression free survival | up to 2 years
  the interval between the time of treatment initiation to the time of progressive disease or patient death
Overall survival | up to 2 years
  the interval between the time of treatment initiation to the time of patient death
Ratio of R0 resection | up to 2 years
  The ratio of patients who underwent R0 resection to patients received combination therapy
Recurrence-free survival | up to 5 years
  the interval between the time of surgical resection to the time of disease recurrence or patient death for those who underwent surgery
Time to deterioration in patient-reported quality of life, physical functioning, and role functioning | up to 2 years
  Quality of life, physical functioning, and role functioning was determined by EORTC QLQ-C30 and QLQ-HCC18 questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Sun, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No